CLINICAL TRIAL: NCT03352284
Title: Replacement of Individual Teeth in the Esthetic Zone of Upper Jaw by Using a Monoblock Ceramic Implant: One Year Follow up
Brief Title: Single Tooth Restoration in the Maxilla Using the Straumann® PURE® Ceramic Implant Monotype: One Year Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miren Vilor Fernández (Other)
Responsible Party: Sponsor-Investigator, Miren Vilor Fernández, Principal Investigator, University of the Basque Country (UPV/EHU)
Organization: University of the Basque Country (UPV/EHU) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017_03
Record Dates: First submitted 2017-11-19; First posted 2017-11-24 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Ceramic Implant
Keywords: Zirconia implant; One-piece; Monoblock; Single tooth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Straumann Pure Ceramic Implant (Experimental): Replacement of single tooth gaps with a Zirconia implant
  Interventions: Device: Straumann Pure Ceramic Implant

INTERVENTIONS:
Device: Straumann Pure Ceramic Implant — The surgical technique begins with the lift of a vestibular mucoperiosteal flap respecting the papillae of the adjacent teeth. After the alveolar bone is exposed, the sequence of drilling and placement of the intra-bone fixation are carried out. In case of fenestrations or dehiscence, they are treated by xenograft and collagen-absorbable membrane. Once the implant is placed, a healing cap or provisional prosthesis is placed depending on the torque achieved. Finally, the flap is replaced and sutured.

SUMMARY:
The main objective is to evaluate peri-implant hard and soft tissues's stability with the use of a ceramic implant (Implant Straumann®Pure Ceramic) during one year follow up.

DETAILED DESCRIPTION:
Nowadays, the material of choice for the manufacture of dental implants is titanium. However, if we consider the aesthetics, the use of metallic implants can lead to complications, namely metal translucency through the peri-implant mucosa or the presence of soft tissue recessions causing metal exposure. As an alternative to the use of titanium, we have zirconium, that is highly biocompatible and whose use in implantology has demonstrated a predictable osseointegration. In addition, some studies suggest a different histology that could help maintaining the stability of the peri-implant mucosa and, therefore, an improvement in long-term aesthetic results.

The reason for designing this study is that there is not too much data about this type of implants, that can be, really, an alternative to those we know.

To achieve those objectives a single-arm clinical trial is designed, using marginal bone loss as a primary response variable. It is estimated with the calculation of the sample size, we would need 30 patients to get relevant data.

An experienced surgeon (M.V) will perform implant surgery. Later, experienced and calibrated examiners (R.E and E.RG) will collect the following clinical parameters at baseline, and at 4, 8 and 12 months: gingival recession, papillary Jemt index, width and height of the keratinized gingiva, probing depth, plaque index and bleeding on probing.

Finally, a blind statistic (X.M) will analyze the data using the SPSS software, having as unit of analysis the implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Master of Periodontology of the UPV/EHU
* Age > 18 years
* Patient with one single tooth gap in the anterior maxilla
* Plaque and bleeding index (FMPS < 20%).
* Treated periodontal conditions
* The patient is able to fully understand the nature of the proposed surgery and is able to provide a signed informed consent

Exclusion Criteria:

* General contraindications for dental and/or surgical treatment are present.
* The patient is taking medications or having treatments which have an effect on healing in general (e.g. steroids, large doses of anti-inflammatory drugs).
* Untreated periodontal conditions
* Patients not willing to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Marginal bone level change (MBLC) | Change from baseline until 12 months
  Distance between the mesial/distal marginal crests and the first implant thread. This is calibrated based on the known length (1,8 mm) of the machined neck.

SECONDARY OUTCOMES:
Gingival recession (REC) | Change from baseline (when the crown is cemented) until 12 months.
  Distance in mm from incisal edge to gingival margin.
Jemt Papilla index score (JPIS) | Change from baseline until 12 months.
  This score ranges from 0 to 3. Index score 0 denotes no soft tissue in the area; index score 1 denotes soft tissue reaching less than half the distance between the reference line and the contact point; index score 2 denotes more soft tissue than indicated by index score 1 but not extending all the way to the contact point; and index score 3 denotes tissue filling the entire embrasure.
Surgical complications (SC) | Surgery and the next 7 days.
  Any complication, as bleeding, dehiscence, loss of suture, etc... that may appear will be collected.
Prosthetic complications (PC) | Baseline, 4, 8 and 12 months.
  Any difficulty during the confection of the crown, complications as descementation, chipping, etc... will be registered.
Probing depth (PD) | Baseline, 4, 8 and 12 months.
  Distance in mm from the gingival margin to the bottom of peri-implant pocket. It will be recorded in 6 points (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual).
Bleeding on probing (BOP) | Baseline, 4, 8 and 12 months.
  Presence or not of bleeding after probing. It will be recorded in 6 points (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual).
Plaque index (PI) | Baseline, 4, 8 and 12 months.
  A plaque developer is used and the presence of plaque is recorded at 6 points per tooth/implant and the percentage of sites with plaque is calculated (O'Leary et al 1972).
Width of keratinized tissue (WKT) | Baseline and 12 months.
  Distance in mm from the mucogingival junction to the gingival margin, measured at the vestibular midpoint.
Thickness of keratinized tissue (TKT) | Baseline and 12 months
  The thickness of the gingiva around the implant is measured approximately 2 mm apical to gingival margin on the facial aspect of the implant. After topical application of anesthetic, the thickness is measured by gently inserting a 27-gauge needle with a rubber stopper in the tip until the underlying hard structure had been contacted. The distance between the tip of the needle and the rubber stopper is measure with a periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Antonio Aguirre Zorzano, Dr., Study Director — University of the Basque Country (UPV/EHU); Luis Barbier Herrero, Dr., Study Director — University of the Basque Country (UPV/EHU); Miren Vilor Fernández, Lcda., Principal Investigator — University of the Basque Country (UPV/EHU); Ana Maria García de la Fuente, Dr., Study Chair — University of the Basque Country (UPV/EHU); Ruth Estefanía Fresco, Dr., Study Chair — University of the Basque Country (UPV/EHU); Xabier Marichalar Mendia, Dr., Study Chair — University of the Basque Country (UPV/EHU); Elena Ruiz de Gopegui Palacios, Lcda., Study Chair — University of the Basque Country (UPV/EHU)
Locations (1):
- Department of Stomatology II, Faculty of Medicine and Nursery, University of the Basque Country, Leioa, Biscay, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gahlert M, Roehling S, Sprecher CM, Kniha H, Milz S, Bormann K. In vivo performance of zirconia and titanium implants: a histomorphometric study in mini pig maxillae. Clin Oral Implants Res. 2012 Mar;23(3):281-6. doi: 10.1111/j.1600-0501.2011.02157.x. Epub 2011 Aug 2. PMID 21806681
- [Background] Kohal RJ, Knauf M, Larsson B, Sahlin H, Butz F. One-piece zirconia oral implants: one-year results from a prospective cohort study. 1. Single tooth replacement. J Clin Periodontol. 2012 Jun;39(6):590-7. doi: 10.1111/j.1600-051X.2012.01876.x. Epub 2012 Apr 23. PMID 22519944
- [Background] Payer M, Arnetzl V, Kirmeier R, Koller M, Arnetzl G, Jakse N. Immediate provisional restoration of single-piece zirconia implants: a prospective case series - results after 24 months of clinical function. Clin Oral Implants Res. 2013 May;24(5):569-75. doi: 10.1111/j.1600-0501.2012.02425.x. Epub 2012 Feb 15. PMID 22335358
- [Background] Gahlert M, Burtscher D, Pfundstein G, Grunert I, Kniha H, Roehling S. Dental zirconia implants up to three years in function: a retrospective clinical study and evaluation of prosthetic restorations and failures. Int J Oral Maxillofac Implants. 2013 May-Jun;28(3):896-904. doi: 10.11607/jomi.2211. PMID 23748325
- [Background] Borgonovo AE, Censi R, Vavassori V, Arnaboldi O, Maiorana C, Re D. Zirconia Implants in Esthetic Areas: 4-Year Follow-Up Evaluation Study. Int J Dent. 2015;2015:415029. doi: 10.1155/2015/415029. Epub 2015 Jun 1. PMID 26124836
- [Background] Gahlert M, Kniha H, Weingart D, Schild S, Gellrich NC, Bormann KH. A prospective clinical study to evaluate the performance of zirconium dioxide dental implants in single-tooth gaps. Clin Oral Implants Res. 2016 Dec;27(12):e176-e184. doi: 10.1111/clr.12598. Epub 2015 Apr 1. PMID 25827600
- [Background] Siddiqi A, Kieser JA, De Silva RK, Thomson WM, Duncan WJ. Soft and Hard Tissue Response to Zirconia versus Titanium One-Piece Implants Placed in Alveolar and Palatal Sites: A Randomized Control Trial. Clin Implant Dent Relat Res. 2015 Jun;17(3):483-96. doi: 10.1111/cid.12159. Epub 2013 Sep 23. PMID 24112624
- [Background] Hashim D, Cionca N, Courvoisier DS, Mombelli A. A systematic review of the clinical survival of zirconia implants. Clin Oral Investig. 2016 Sep;20(7):1403-17. doi: 10.1007/s00784-016-1853-9. Epub 2016 May 24. PMID 27217032
- [Background] Linares A, Grize L, Munoz F, Pippenger BE, Dard M, Domken O, Blanco-Carrion J. Histological assessment of hard and soft tissues surrounding a novel ceramic implant: a pilot study in the minipig. J Clin Periodontol. 2016 Jun;43(6):538-46. doi: 10.1111/jcpe.12543. Epub 2016 May 2. PMID 26969899
- [Background] Gahlert M, Rohling S, Wieland M, Eichhorn S, Kuchenhoff H, Kniha H. A comparison study of the osseointegration of zirconia and titanium dental implants. A biomechanical evaluation in the maxilla of pigs. Clin Implant Dent Relat Res. 2010 Dec;12(4):297-305. doi: 10.1111/j.1708-8208.2009.00168.x. PMID 19438936
- [Background] Oliva J, Oliva X, Oliva JD. Five-year success rate of 831 consecutively placed Zirconia dental implants in humans: a comparison of three different rough surfaces. Int J Oral Maxillofac Implants. 2010 Mar-Apr;25(2):336-44. PMID 20369093
- [Background] Sicilia A, Cuesta S, Coma G, Arregui I, Guisasola C, Ruiz E, Maestro A. Titanium allergy in dental implant patients: a clinical study on 1500 consecutive patients. Clin Oral Implants Res. 2008 Aug;19(8):823-35. doi: 10.1111/j.1600-0501.2008.01544.x. PMID 18705814
- [Background] Grassi FR, Capogreco M, Consonni D, Bilardi G, Buti J, Kalemaj Z. Immediate occlusal loading of one-piece zirconia implants: five-year radiographic and clinical evaluation. Int J Oral Maxillofac Implants. 2015 May-Jun;30(3):671-80. doi: 10.11607/jomi.3831. PMID 26009919
- [Background] Thoma DS, Benic GI, Munoz F, Kohal R, Sanz Martin I, Cantalapiedra AG, Hammerle CH, Jung RE. Marginal bone-level alterations of loaded zirconia and titanium dental implants: an experimental study in the dog mandible. Clin Oral Implants Res. 2016 Apr;27(4):412-20. doi: 10.1111/clr.12595. Epub 2015 Apr 10. PMID 25864523